CLINICAL TRIAL: NCT02651467
Title: A Clinical Study Investigating the Efficacy of Two Experimental Oral Rinses in Providing Long Term Relief From Dentinal Hypersensitivity
Brief Title: A Study to Investigate Efficacy of Two Experimental Oral Rinses in Providing Long Term Relief From Pain Derived From Exposed Dentine in Response to Chemical, Thermal, Tactile, or Osmotic Stimuli.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204763
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Oral Rinse 1 (1.5% w/w KOX, 0ppm F, pH 7.0) (Experimental): Participants will apply a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brush their teeth for one timed minute and expectorate. They will then rinse with 20ml of tap water (using the dosing cap provided) for 10 seconds and expectorate, then rinse with 10ml of the experimental oral rinse 1 (using the second dosing cap provided) for one timed minute and expectorate. No further rinsing will be allowed. This regimen will be performed twice daily for 8 weeks.
  Interventions: Other: Experimental Oral Rinse 1 (1.5% w/w KOX, 0ppm F, pH 7.0)
- Experimental Oral Rinse 2 (2.0% w/w KOX, 45ppm F, pH 4.5) (Experimental): Participants will apply a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brush their teeth for one timed minute and expectorate. They will then rinse with 20ml of tap water (using the dosing cap provided) for 10 seconds and expectorate, then rinse with 10ml of the experimental oral rinse 2 (using the second dosing cap provided) for one timed minute and expectorate. No further rinsing will be allowed. This regimen will be performed twice daily for 8 weeks.
  Interventions: Other: Experimental Oral Rinse 2 (2.0% w/w KOX, 45ppm F, pH 4.5)
- Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ) (Placebo Comparator): Participants will apply a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brush their teeth for one timed minute and expectorate. They will then rinse with 20ml of tap water (using the dosing cap provided) for 10 seconds and expectorate, then rinse with 10ml of the placebo oral rinse (using the second dosing cap provided) for one timed minute and expectorate. No further rinsing will be allowed. This regimen will be performed twice daily for 8 weeks.
  Interventions: Other: Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )

INTERVENTIONS:
Other: Experimental Oral Rinse 1 (1.5% w/w KOX, 0ppm F, pH 7.0) — 1.5% w/w KOX, 0ppm F, pH 7.0
  Arms: Experimental Oral Rinse 1 (1.5% w/w KOX, 0ppm F, pH 7.0)
Other: Experimental Oral Rinse 2 (2.0% w/w KOX, 45ppm F, pH 4.5) — 2.0% w/w KOX, 45ppm F, pH 4.5
  Arms: Experimental Oral Rinse 2 (2.0% w/w KOX, 45ppm F, pH 4.5)
Other: Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ) — 0% w/w KOX 0ppm F, pH 4.5
  Arms: Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )

SUMMARY:
This will be a single center, eight week, randomized, double blind, three treatment arm, parallel design, stratified (by mean baseline Schiff Sensitivity Score of the two selected test teeth) study in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Participants will be male or female aged between 18 and 65 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee.

No clinically significant and relevant abnormalities in medical history or upon oral examination.

Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

* Self-reported history of dentinal hypersensitivity (DH) lasting more than(>) six months but not > 10 years.
* Good general oral health, with a minimum of 20 natural teeth.
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants at screening and minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars) at baseline.

Exclusion Criteria:

* Women who are pregnant or breast-feeding .
* Daily doses of medication/treatments which, in the opinion of the Investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs.
* Currently taking antibiotics or has taken antibiotics within two weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Presence of kidney disease, hyperoxaluria, or any other condition that may be exacerbated by oxalic acid or oxalate salts.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* Dental prophylaxis within four weeks of Screening, tongue or lip piercing or presence of dental implants.
* Desensitizing treatment within eight weeks of Screening (professional sensitivity treatments and non-toothpaste sensitivity treatments).
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within eight weeks of Screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter toothpaste in the opinion of the Investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within eight weeks of screening.
* Individuals who require antibiotic prophylaxis for dental procedures.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-01-04; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in USA.
Pre-assignment Details: Total 265 participants were screened, out of which 221 participants were randomized. 44 participants were not randomized; 43 participants did not meet the study criteria and 1 participant withdraw his consent before getting randomized to any study treatment.
Groups:
- Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20millilitre (mL) of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Treatment 1 (Oral rinse 1.5% weight by weight [w/w] KOX, 0 parts per million [ppm], pH 7.0) (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
- Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Treatment 2 (Oral rinse 2.0% w/w KOX, 45ppm F, pH 4.5) (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
- Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ) (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
Started | 74 | 74 | 73
Completed | 73 | 74 | 69
Not Completed | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Other (Not specified) | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all the participants who were randomized and received at least one dose of study treatment during the study.
Groups:
- Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Treatment 1 (Oral rinse 1.5% w/w KOX, 0ppm F, pH 7.0) (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ) | Total
Number analyzed (Participants) | 74 | 74 | 73 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (12.41) | 44.9 (11.99) | 44.4 (12.33) | 44.4 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 64 | 184
  Male | 14 | 14 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 8 (Treatment 1 and 2 Versus [vs.] Placebo)
Description: Schiff sensitivity score was assessed by participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth, response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Time Frame: Baseline and Week 8
Population: Intent-to-treat (ITT) population (N=218), defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy. This analysis was conducted on ITT population. Baseline data only includes those participants who have a corresponding post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
Number analyzed (Participants) | 74 | 74 | 70
Score on scale
  Schiff score at baseline: number analyzed (Participants) | 73 | 74 | 69
  Schiff score at baseline | 2.51 (0.408) | 2.53 (0.408) | 2.54 (0.409)
  Change from baseline in Schiff score at Week 8: number analyzed (Participants) | 73 | 74 | 69
  Change from baseline in Schiff score at Week 8 | -1.57 (0.756) | -1.72 (0.764) | -0.69 (0.875)
Statistical Analysis 1: Comparison: Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) vs Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ); For the Week 8 comparisons of the two Treatments against the Placebo Control, Dunnett's multiplicity adjustment is applied; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = -0.88, 95% CI 2-sided [-1.181 to -0.584] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) vs Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ); For the Week 8 comparisons of the two Treatments against the control, Dunnett's multiplicity adjustment is applied; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Diference of Least Square mean = -1.04, 95% CI 2-sided [-1.333 to -0.738] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 8 (Treatment 1 vs. Treatment 2)
Description: as for outcome 1
Time Frame: Baseline and Week 8
Population: Intent-to-treat (ITT) population (N=218), defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy. Data shown for Treatment 1& 2 only for this endpoint. Baseline data only includes those participants who have a corresponding post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5)
Number analyzed (Participants) | 74 | 74
Score on a scale
  Schiff score at Baseline: number analyzed (Participants) | 73 | 74
  Schiff score at Baseline | 2.51 (0.408) | 2.53 (0.408)
  Change from baseline in Schiff score at Week 8: number analyzed (Participants) | 73 | 74
  Change from baseline in Schiff score at Week 8 | -1.57 (0.756) | -1.72 (0.764)
Statistical Analysis 1: Comparison: Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) vs Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5); Test type: Superiority or Other; p = 0.2478, ANCOVA — From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Least Square Mean Difference = 0.15, 95% CI [-0.107 to 0.413] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Week 4
Description: Schiff sensitivity score was assessed as participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth, using scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of syimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3=Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Time Frame: Baseline and Week 4
Population: Intent-to-treat (ITT) population (N=218), defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
Number analyzed (Participants) | 74 | 74 | 70
Score on scale
  Shiff score at baseline | 2.52 (0.409) | 2.53 (0.408) | 2.54 (0.411)
  Change from baseline in Schiff score at Week 4 | -1.04 (0.814) | -1.18 (0.846) | -0.50 (0.761)

4. Secondary Outcome: Change From Baseline in Tactile Threshold at Week 4 and 8
Description: Pressure was administered using a constant pressure probe (Yeaple Probe). The constant pressure probe allows the examiner to vary the force applied to the dentine surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline, Week 4 and 8
Population: Intent-to-treat (ITT) population (N=218), defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
  Note: Baseline population only includes those subjects who have a corresponding post-baseline assessment.
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )(using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
Number analyzed (Participants) | 74 | 74 | 70
grams
  Tactile threshold at baseline for Week 4 | 10.14 (0.816) | 10.14 (0.816) | 10.00 (0.000)
  Change at Week 4 | 37.91 (26.276) | 47.16 (26.133) | 15.29 (23.558)
  Tactile threshold at baseline for Week 8: number analyzed (Participants) | 73 | 74 | 69
  Tactile threshold at baseline for Week 8 | 10.14 (0.822) | 10.14 (0.816) | 10.00 (0.000)
  Change at Week 8: number analyzed (Participants) | 73 | 74 | 69
  Change at Week 8 | 53.56 (21.024) | 57.91 (25.062) | 17.39 (28.743)

5. Secondary Outcome: Change From Baseline in Visual Rating Scale (VRS) at Week 4 and 8
Description: Participants rated the intensity of their response to the evaporative (air) stimulus using a 10 point VRS. The subjects were asked to rate their pain on a scale of 1 ("No Pain") to 10 ("Intense Pain").
Time Frame: Baseline, Week 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
Number analyzed (Participants) | 74 | 74 | 70
Score on a scale
  VRS at baseline for Week 4 | 6.56 (1.969) | 6.55 (1.952) | 6.60 (1.777)
  VRS at Week 4 | -2.05 (1.805) | -2.09 (1.675) | -1.46 (1.862)
  VRS at baseline for Week 8: number analyzed (Participants) | 73 | 74 | 69
  VRS at baseline for Week 8 | 6.55 (1.982) | 6.55 (1.952) | 6.64 (1.749)
  VRS at Week 8: number analyzed (Participants) | 73 | 74 | 69
  VRS at Week 8 | -3.13 (2.012) | -3.34 (1.756) | -2.27 (2.105)

ADVERSE EVENTS:
Groups:
- Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20millilitre (mL) of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Treatment 1 (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
- Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Treatment 2 (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
- Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ): Participants applied a strip of standard fluoride toothpaste to cover the full head of the toothbrush and brushed their teeth for one timed minute and expectorated. After that, they rinsed with 20mL of tap water (using the dosing cap provided) for 10 seconds and expectorated, then again rinsed with 10mL of Placebo oral rinse (using the second dosing cap provided) for one timed minute and expectorated. No further rinsing was allowed. This regimen was performed twice daily for 8 weeks.
Arm/Group | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 )
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 4/74 | 2/74 | 5/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 (Oral Rinse 1.5% w/w KOX, 0ppm F, pH 7.0) (N=74) | Treatment 2 (Oral Rinse 2.0% w/w KOX, 45ppm F, pH 4.5) (N=74) | Placebo Oral Rinse (0% w/w KOX 0ppm F, pH 4.5 ) (N=73)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0 (0) | 2
OEDEMA MOUTH (Gastrointestinal disorders) | 0 (0) | 1 | 0 (0)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1
LIP ULCERATION (Gastrointestinal disorders) | 1 | 0 (0) | 0
BURN ORAL CAVITY (Injury, poisoning and procedural complications) | 1 | 1 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.